CLINICAL TRIAL: NCT02136693
Title: Efficacia Della Fibra di Psyllium Versus Placebo Nella Gestione Dell'Alvo in Pazienti Sottoposti ad Intervento Chirurgico Per Ostruita Defecazione
Brief Title: Psyllium Fiber Versus Placebo in Early Treatment After STARR for Obstructed Defecation: a Double-blind RCT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Francesco Gabrielli (Other)
Responsible Party: Sponsor-Investigator, Francesco Gabrielli, professore ordinario di chirurgia generale, University of Milano Bicocca
Organization: University of Milano Bicocca (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: psyllium_STARR
Record Dates: First submitted 2014-05-05; First posted 2014-05-13 (Estimated); Last update posted 2014-05-13 (Estimated); Status verified 2014-05

CONDITIONS: Constipation; Incontinence
Keywords: obstructed defecation; STARR; constipation; incontinence; psyllium
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): 3.5 g /day of inert compound for 180 days after STARR
  Interventions: Drug: Placebo
- Psyllium fiber (Experimental): 3.5 g /day of pure Psyllium fiber for 180 days after STARR
  Interventions: Drug: Psyllium fiber

INTERVENTIONS:
Drug: Psyllium fiber — 3.5 g /day of pure Psyllium fiber for 180 days after STARR
  Arms: Psyllium fiber
Drug: Placebo — 3.5 g /day of inert compound for 180 days after STARR
  Other Names: inert compound
  Arms: Placebo

SUMMARY:
This study aims to assess whether fiber intake, formerly recommended only before or instead of surgery, may play a role in improving postoperative progress and functional outcome after STARR for obstructed defecation, in terms of residual constipation, incontinence and defecation urgency.

DETAILED DESCRIPTION:
After obtaining written informed consent and collecting baseline scores (T0), each patient was randomly assigned to one of the two groups and began taking sachets containing Psyllium fiber 3.5 g / day for Active group (A) and inert compound for Placebo group (P).

Sachet content was assigned by software randomization, written on a list and sealed in an envelope, which was opened only after the study was completed.

Post-operative instructions for both groups included only analgesic therapy (Ketorolac 10 to 30 mg b.m. if needed). Patients were also asked to stop any former laxative and to continue on a normal diet.

Each patient was re-evaluated at 7 ± 3 (T1), 60 ± 5 (T2) and 180 ± 15 (T3) days after surgery (Table 2).

A fluoroscopic colpocystodefecography (with patient sitting upright) was obtained before surgery and between 60-180 days postoperatively in order to assess comparability of the two groups and exclude negative organic outcomes that could affect functional results.

Medical events were investigated while checking each patient, with special regard to defecation urgency. From the data collected on concomitant medications, we extrapolated those related to laxative intake.

The treatment was considered accomplished in patients who had taken at least 70% of the product during each interval of follow-up.

Statistical analysis was performed using the SPSS - PASW Statistics 18.0.0 (IBM ©, 2009).

For the general and defecographic characteristics, the data are expressed in the form of mean ± standard deviation for continuous variables and absolute frequency (frequency percentages) for categorical variables. The differences between the two groups were calculated by two-tailed t-test or chi-square when appropriate.

Scores for the assessment of clinical data are expressed as mean ± standard deviation and analysis of the differences in the two groups was performed using the two-tailed t-test. The analysis of not normally distributed variables was conducted using a non-parametric test (Wilcoxon-Mann-Whitney).

Analyses related to defecation urgency and use of laxatives were carried out using chi-square test and the data are expressed as absolute frequency (frequency percentage).

For all tests, a value of p <0.05 was considered significant.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Age over 18
* Diagnosis of Obstructed Defecation Syndrome according to ODS and CCS Score
* STARR performed when ODS score >10
* STARR performed 48-72 hours before

Exclusion Criteria:

* Puborectalis or sphincter dyssynergia, evaluated by defecography and / or anorectal manometry
* Concomitant diseases (fissure, abscess, fistula, IBD, diverticular disease)
* Prolapse of other pelvic floor organs
* Proctological surgery before STARR
* Pregnancy or breast-feeding
* Ongoing treatment with oral anticoagulants or steroid therapy
* Conditions that do not allow patients to understand the nature and the purpose of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2010-05; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
residual constipation | 180 days after STARR
  ODS score and CCS score

SECONDARY OUTCOMES:
Post-operative pain | 180 days after STARR
  VAS
revertence to laxative use | 180 days after STARR
  frequency percentage of patients that reverted to laxative use after surgery
change in fecal incontinence from baseline | 180 days after STARR
  Wexner Incontinence score
post-operative defecation urgency | 180 days after STARR
  defecation urgency incidence

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Gabrielli, Prof., Study Chair — Università degli studi Milano Bicocca
Locations (1):
- Istituti Clinici Zucchi, Monza, MB, Italy